CLINICAL TRIAL: NCT02095340
Title: Effects of Maternal Interpretation Biases on Child Anxiety and Related Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Andres G. Viana, Assistant Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014-0035
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Training (Experimental)
  Interventions: Other: Positive Interpretation Bias Training
- Neutral Training (Sham Comparator)
  Interventions: Other: Neutral Interpretation Bias Training

INTERVENTIONS:
Other: Positive Interpretation Bias Training
  Arms: Positive Training
Other: Neutral Interpretation Bias Training
  Arms: Neutral Training

SUMMARY:
The purpose of this study is to expand our understanding of the intergenerational transmission of cognitive risk for childhood anxiety disorders by examining whether changes in maternal interpretations of situations result in changes in child interpretations and child anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-12
* Children with primary diagnosis of anxiety disorder
* Mothers with clinical levels of anxiety symptoms on the Depression, Anxiety, and Stress Scales (DASS; Lovibond & Lovibond, 1995)

Exclusion Criteria:

* Physical disability impairing ability to use a computer
* Intelligence Quotient <80
* Reading comprehension and fluency composite <75
* Concurrent primary diagnosis of any non-anxiety disorder
* Currently receiving psychological or pharmacological treatment for anxiety
* Danger to self/others
* Non-English speaking child/parent
* Maternal current involvement in cognitive-behavioral therapy
* Maternal changes in pharmacological treatment in the 12 weeks prior to enrollment.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2014-05; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Raines EM, Viana AG, Trent ES, Conroy HE, Woodward EC, Zvolensky MJ, Storch EA. The explanatory role of anxiety sensitivity in the association between effortful control and child anxiety and depressive symptoms. Cogn Behav Ther. 2020 Nov;49(6):501-517. doi: 10.1080/16506073.2020.1790644. Epub 2020 Jul 21. PMID 32692282
- [Derived] Trent ES, Viana AG, Raines EM, Conroy HE, Storch EA, Zvolensky MJ. Interpretation biases and depressive symptoms among anxiety-disordered children: The role of individual differences in respiratory sinus arrhythmia. Dev Psychobiol. 2021 Mar;63(2):320-337. doi: 10.1002/dev.22002. Epub 2020 Jun 10. PMID 32524580
- [Derived] Trent ES, Viana AG, Raines EM, Woodward EC, Candelari AE, Storch EA, Zvolensky MJ. Interpretation Biases and Childhood Anxiety: The Moderating Role of Parasympathetic Nervous System Reactivity. J Abnorm Child Psychol. 2020 Mar;48(3):419-433. doi: 10.1007/s10802-019-00605-7. PMID 31802369
- [Derived] Raines EM, Viana AG, Trent ES, Woodward EC, Candelari AE, Zvolensky MJ, Storch EA. Effortful control, interpretation biases, and child anxiety symptom severity in a sample of children with anxiety disorders. J Anxiety Disord. 2019 Oct;67:102136. doi: 10.1016/j.janxdis.2019.102136. Epub 2019 Aug 27. PMID 31494512

RESULTS

PARTICIPANT FLOW:
Groups:
- Positive Training: Positive Interpretation Bias Training
- Neutral Training: Neutral Interpretation Bias Training
- Child Interpretation Biases Assessment: All children, regardless of whether the parent was assigned to either the positive or neutral training condition, completed a single assessment of interpretation biases.
Period: Overall Study
Arm/Group | Positive Training | Neutral Training | Child Interpretation Biases Assessment
Started | 51 (Mother (not the child) received the training.) | 54 (Mother (not the child) received the training.) | 105
Completed | 51 | 54 | 105
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Training | Neutral Training | Child Interpretation Biases Assessment | Total
Number analyzed (Participants) | 51 | 54 | 105 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 105 | 105
  Between 18 and 65 years | 51 | 54 | 0 | 105
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.73 (6.92) | 39.94 (7.19) | 10.07 (1.22) | 29.58 (5.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 54 | 60 | 165
  Male | 0 | 0 | 45 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 13 | 18 | 30 | 61
  African American | 7 | 8 | 15 | 30
  White American | 27 | 27 | 40 | 94
  Asian American | 2 | 0 | 2 | 4
  Mixed Ethnicity | 2 | 1 | 18 | 21
Region of Enrollment [Number; unit: participants]
  United States | 51 | 54 | 105 | 210
Word-Sentence Association Paradigm [Mean (Standard Deviation); unit: Units on a Scale] — Proportion of threatening vs non-threatening interpretations made on the modified version of the Word Sentence Association Paradigm (WSAP). Score ranges from 0 to 1. Higher scores indicate worse outcome, that is, more negative interpretation biases.
  Units on a Scale | 0.53 (0.14) | 0.52 (0.12) | 0.27 (0.15) | 0.44 (0.14)

OUTCOME MEASURES:

1. Primary Outcome: Word Sentence Association Paradigm
Description: Proportion of threatening (versus nonthreatening) interpretations made on the Word Sentence Association Paradigm (WSAP). Scores range from 0 to 1. Higher scores mean a worse outcome, that is, more negative interpretations.
Time Frame: Participants will be assessed, on average, within 20 minutes after the intervention.
Population: Data for one participant in the positive training condition and two participants in the neutral training condition was lost due to equipment malfunction.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Child Interpretation Biases Assessment: All children completed a Child Interpretation Biases Assessment once.
Arm/Group | Positive Training | Neutral Training | Child Interpretation Biases Assessment
Number analyzed (Participants) | 50 | 52 | 105
units on a scale | 0.37 (0.16) | 0.52 (0.14) | 0.27 (0.15)

2. Primary Outcome: Maternal Anxious Behavior Coded by Independent Observers.
Description: Maternal anxious behavior coded by independent observers on a 0 - 4 scale. Higher numbers indicated more observed anxious behaviors.
Time Frame: Immediately after the intervention, an average of 10 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Child Interpretation Biases Assessment: Child Interpretation Biases Assessment
Arm/Group | Positive Training | Neutral Training | Child Interpretation Biases Assessment
Number analyzed (Participants) | 51 | 54 | 105
units on a scale | 1.43 (0.81) | 1.70 (0.79) | 2.02 (0.93)

ADVERSE EVENTS:
Time Frame: The day of the intervention.
Description: There were no adverse events or serious adverse events during the trial. All-Cause Mortality was not monitored/assessed and therefore the total number of participants at risk is listed as zero ("0").
Arm/Group | Positive Training | Neutral Training | Child Interpretation Biases Assessment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/54 | 0/105
Other Adverse Events (participants affected / at risk) | 0/51 | 0/54 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT02095340/Prot_SAP_000.pdf